CLINICAL TRIAL: NCT02902276
Title: Link Between Plasma Citrulline and Lipopolysaccharide Concentrations in the Critically Ill
Acronym: CITRANS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2016/187
Record Dates: First submitted 2016-08-11; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Critically Ill
Keywords: plasma citrulline; lipopolysaccharide; critically ill; Hospitalization in an Intensive Care Unit
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2000 microliters of plasma will be stored at -80°C for future analyses (lipopolysaccharide concentration, cytokines).
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: additional blood sample — Two blood samples will be taken at ICU admission

SUMMARY:
In critically ill patients, the small bowel permeability is increased, leading to bacterial translocation, and systemic inflammatory response syndrome.

Plasma citrulline is a validated biomarker of functional enterocyte mass. Lipopolysaccharide (LPS) is a part of Gram negative bacteria, and plasma LPS concentration is a biomarker of bacterial translocation. The link between plasma citrulline and LPS in the critically ill is unknown. Investigators hypothesize that patients presenting with low plasma citrulline concentration, with presumed altered small bowel function, would have an increased phenomenon of bacterial translocation, and increased plasma LPS concentration. Investigators aimed to evaluate the link between plasma citrulline and LPS concentrations in critically ill patients at the time of ICU admission.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients requiring ICU admission for at least 48 hours
* Adults

Exclusion Criteria:

* Chronic small bowel disease
* Chronic renal failure (clearance of creatinine < 50 mL/min)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients requiring ICU admission for at least 48 hours, without chronic small bowel disease, without chronic renal failure (usual clearance of creatinine < 50 mL/min), not pregnant.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Plasma citrulline concentration | Up to 12 hours after admission in the unit
  biological assay
plasma lipopolysaccharide concentration | Up to 12 hours after admission in the unit
  biological assay

CONTACTS AND LOCATIONS:
Overall Officials: Gaël Piton, MD, PhD, Principal Investigator — CHU Besançon
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chaignat C, Lagrost L, Moretto K, de Barros JP, Winiszewski H, Grober J, Saas P, Piton G. Plasma citrulline concentration and plasma LPS detection among critically ill patients a prospective observational study. J Crit Care. 2024 Feb;79:154438. doi: 10.1016/j.jcrc.2023.154438. Epub 2023 Oct 3. PMID 37797404